CLINICAL TRIAL: NCT05481411
Title: A Phase I, Open-label Single Dose Study to Evaluate the Pharmacokinetics, Safety, and Pharmacodynamics of Olpasiran in Subjects With Various Degrees of Hepatic Impairment
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Pharmacodynamics of Olpasiran in Participants With Various Degrees of Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20220009
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Hepatic Impairment
Keywords: Olpasiran; Hepatic Impairment; Normal Hepatic Function; AMG 890
MeSH Terms: interventions — olpasiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Dose Olpasiran Hepatic Impairment (Experimental): Participants will be enrolled in 1 of 3 hepatic impairment groups based on their hepatic impairment status, as determined by Child-Pugh classification. All participants will receive a single dose of olpasiran on Day 1.
  Interventions: Drug: Olpasiran
- Single Dose Olpasiran Normal Hepatic Function (Experimental): Participants with normal hepatic function will be enrolled and will receive a single dose of olpasiran on Day 1.
  Interventions: Drug: Olpasiran

INTERVENTIONS:
Drug: Olpasiran — Subcutaneous injection
  Other Names: AMG 890

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetics (PK) of a single dose of olpasiran in participants with mild, moderate, or severe hepatic impairment compared to participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants of nonchildbearing potential, between 18 and 75 years of age (inclusive) at the time of Screening.
* Body mass index between 18.0 and 40.0 kg/m^2 (inclusive) at the time of Screening.

Participants with Normal Hepatic Function Only:

• In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations at Screening and Check-in as assessed by the Investigator (or designee).

Participants with Hepatic Impairment Only:

• Child-Pugh A (Group 2), B (Group 3), or C (Group 4) classification defined by both Screening (to determine participant group) and Check-in (to confirm participant group prior to dosing) clinical laboratory values and physical examination findings.

Exclusion Criteria:

* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
* Estimated glomerular filtration rate < 60 mL/min/1.73m^2 (Groups 1-3) or < 50 mL/min/1.73m^2 (Group 4 only) by Modification of Diet in Renal Disease formula at Screening or Check-in.
* Receiving or has received any investigational drug within the 30 days or 5 half-lives (whichever is longer) before receiving olpasiran.
* Participants who were previously exposed to olpasiran.
* Female participants with a positive pregnancy test at Screening or Check-in.

Participants with Normal Hepatic Function Only:

* Positive hepatitis panel. Participants whose results are compatible with prior immunization may be included.
* Alanine aminotransferase and aspartate aminotransferase elevations > 3x upper limit of normal at Screening or Check-in.

Participants with Hepatic Impairment Only:

* Positive for hepatitis B surface antigen. Participants with positive hepatitis B core antibody may be included if hepatitis B surface antigen is negative. Participants with positive hepatitis B surface antibody may be included (consistent with prior vaccination).
* Active malignancy of any type. Participants with a history of malignancy that has been eradicated with supporting medical documentation indicating that there is no residual malignancy detected in the past 2 years will be allowed.
* Values outside the normal range for liver function tests that are not consistent with their hepatic condition, as determined by the Investigator (or designee).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of Olpasiran | Predose, 0.5, 1, 3, 6, 9, 12, 24, 36, 48, 72, 96, 144 hours (postdose), Day 15, and Day 29
Area Under the Plasma Concentration-time Curve from Time Zero to the Last Quantifiable Concentration (AUClast) of Olpasiran | Predose, 0.5, 1, 3, 6, 9, 12, 24, 36, 48, 72, 96, 144 hours (postdose), Day 15, and Day 29
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Olpasiran | Predose, 0.5, 1, 3, 6, 9, 12, 24, 36, 48, 72, 96, 144 hours (postdose), Day 15, and Day 29

SECONDARY OUTCOMES:
Area Under the Effect Time Curve (AUEC) of Plasma Lipoprotein a (Lp[a]) | Screening, Day 1, Day 2, Day 4, Day 7, Day 15, Day 29, Day 57, and Day 85
Maximum Inhibitory Effect (Imax) of Plasma Lp(a) | Screening, Day 1, Day 2, Day 4, Day 7, Day 15, Day 29, Day 57, and Day 85
Time to Reach Imax of Lp(a) | Screening, Day 1, Day 2, Day 4, Day 7, Day 15, Day 29, Day 57, and Day 85
Number of Participants Who Experience an Adverse Event (AE) | Up to Day 85
Number of Participants with Clinically Significant Changes in Clinical Laboratory Evaluations | Up to Day 85
Number of Participants With Clinically Significant Changes 12-lead Electrocardiogram (ECG) Measurements | Up to Day 85
Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Orlando Clinical Research Center, Orlando, Florida
  - The Texas Liver Institute, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com